CLINICAL TRIAL: NCT03780764
Title: Changes in Pulpal Blood Flow of Teeth During Leveling and Alignment Stages of Orthodontic Treatment Using 2 Fixed Orthodontic Appliances
Brief Title: Changes in Pulpal Blood Flow Between Conventional and Self-ligating Fixed Orthodontic Brackets During Leveling and Alignment Stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Proffessor- Main investigator, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 236/2016
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Orthodontic Appliances
Keywords: Pulpal blood flow; self ligating brackets; orthodontics

STUDY DESIGN:
Intervention Model Description: A split mouth study design was applied for each patient. Two different fixed appliance brackets were used in the lower arch (self-ligating brackets on one side and conventional brackets on the other side of the same patients).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional fixed appliance (Active Comparator): A pre-adjusted edgewise fixed appliance (3M Gemini Unitek, 0.022" Roth prescription brackets) on one side of lower arch.
  Interventions: Other: A Pre-adjusted edgewise brackets: 3M Gemini Unitek, 0.022" Roth prescription brackets
- Self ligating fixed appliance (Experimental): Self-ligating brackets (Unitek™ Gemini SL Self-Ligating Brackets, 0.022" Roth prescription brackets) on the other side.
  Interventions: Other: Self- ligating brackets: Unitek™ Gemini SL Self-Ligating Brackets, 0.022" Roth prescription brackets

INTERVENTIONS:
Other: A Pre-adjusted edgewise brackets: 3M Gemini Unitek, 0.022" Roth prescription brackets — A pre-adjusted edgewise fixed appliance (3M Gemini Unitek, 0.022" Roth prescription brackets) on one side of lower arch. The standardized bonding technique was applied according to the manufacturer's instructions. Teeth alignment was initiated using round 0.016" NiTi arch wire until 0.016X0.022" NiTi was reached. The NiTi arch wires were placed into brackets slots and tied with elastomers (figure of 8).
  Arms: Conventional fixed appliance
Other: Self- ligating brackets: Unitek™ Gemini SL Self-Ligating Brackets, 0.022" Roth prescription brackets — Self-ligating brackets (Unitek™ Gemini SL Self-Ligating Brackets, 0.022" Roth prescription brackets) on the other side of lower arch. The standardized bonding technique was applied according to the manufacturer's instructions. Teeth alignment was initiated using round 0.016" NiTi arch wire until 0.016X0.022" NiTi was reached. The NiTi arch wires were placed into brackets slots and held in place by bracket's gate in the self-ligating brackets side.
  Arms: Self ligating fixed appliance

SUMMARY:
- Evaluate and compare initial changes in PBF between conventional and self-ligating fixed orthodontic brackets during leveling and alignment stage using 0.016" Nickle titanium (NiTi) and 0.016X0.022" NiTi archwires at different time intervals (20min, 24h, 72h, 1 week and 1 month) of initial arch wire placement.

DETAILED DESCRIPTION:
Objectives: to evaluate and compare the initial changes in pulpal blood flow (PBF) between conventional and self-ligating fixed orthodontic brackets during leveling and alignment stage.

Materials and Methods: A total of 22 patients (16 females and 6 males) aged 19± 2.53 years who presented with mild lower arch crowding were selected to participate in the study. A split mouth study design was applied for each patient. Two different fixed appliance brackets were used in the lower arch (self-ligating brackets on one side and conventional brackets on the other side of the same patients). PBF was measured for the lower right and left sides using Laser Doppler Flowmetry at different time intervals (20min, 24h, 72h, 1 week and 1 month) after the fitting of 2 alignment archwires; 0.016" NiTi and 0.016X0.022" NiTi. A repeated measures analysis of variance test and a Bonferroni post-hoc comparison test were applied to detect differences in PBF between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects
* 6 or more years old
* Class I skeletal malocclusion
* mild lower arch crowding.

Exclusion Criteria:

* Poor oral hygiene
* Previous orthodontic treatment
* Active periodontal disease
* Missing teeth, deep carious teeth
* Teeth with root resorption
* Endodontically treated teeth
* History of previous trauma
* Restoration on measured teeth
* Medical conditions affecting blood vessels and
* smoking

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Pulpal blood flow changes by the use of Laser Doppler Flowmeter | 20 minutes ,48 hours, 72 hours and 1 month
  millimeter per second

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of science and technology Dental Teaching Clinics, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided